CLINICAL TRIAL: NCT00370188
Title: Clinical Assessment of Topiramate on Gambling-Related Behaviours in Problem Gamblers: Effects of Gender and Negative Emotionality
Brief Title: Topiramate on Gambling-Related Behaviours
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change to investigator's research affiliation and other employment.
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bruna Brands, Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96/2006
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Gambling
Keywords: problem gambling; topiramate
MeSH Terms: conditions — Gambling | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The quest for an effective medication therapy for problem gambling remains an important priority for the problem gambling treatment research field. While several medications have been evaluated in controlled clinical trials, no medication has been shown to unequivocally reduce gambling behaviour and, to date, no medication has been approved for treating this disorder. Recently, topiramate, indicated for the treatment of seizure disorders, has shown some promise as a medication therapy for problem gambling. In this project, the efficacy of topiramate will be evaluated in a placebo-controlled clinical trial, the first study to do so. The interaction of the effects of the medication and gambling sub-type will be examined to determine whether the efficacy of topiramate is correlated with the specific biopsychosocial history of the gambler.

DETAILED DESCRIPTION:
The quest for an effective pharmacotherapy for problem gambling remains an important priority for the problem gambling treatment research field. While several medications have been evaluated in controlled clinical trials no medication has been shown to unequivocally reduce gambling behaviour and, to date, no medication has been approved for treating this disorder. Recently, topiramate, indicated for the treatment of seizure disorders, has shown some promise as a pharmacotherapy for problem gambling. The most persuasive evidence for the efficacy of topiramate has been reported for alcohol (in a placebo-controlled study) and for problem gambling (in which fluvoxamine served as an active control). No study has examined the efficacy of topiramate in a placebo-controlled clinical trial or examined its efficacy within specific sub-groups of gamblers.

Topiramate has recently been found to be effective in a number of psychiatric and addictive disorders. Dannon reported the first trial evaluating topiramate as a treatment for pathological gambling, comparing it to fluvoxamine. Treatment was delivered over a 12-week period with a maximum dose of 200 mg/d. Nine out of 15 topiramate subjects had achieved full remission of gambling behaviour compared to 6 out of 16 fluvoxamine subjects. However, both groups improved to a similar degree on other measures of psychopathology (e.g., anxiety). This study and Dannon's previous study of topiramate's efficacy in the treatment of kleptomania, suggests that topiramate may be particularly effective for Impulse-Control Disorders.

Topiramate-induced modulation of the noradrenergic pathways that mediate hyper- arousal, conditionability and intrusive/ emotional memories suggests that this medication may be particularly efficacious in problem gamblers characterized by hyper-arousal, anxiety and depression. Blaszczynski in their delineation of the Pathways Model of problem and pathological gambling, has identified a group of problem gamblers who self-regulate dysphoric emotional states through escape, dissociation and numbing (i.e., Emotionally Vulnerable problem gamblers). The Impulsivist and the Conditioned problem gambler, the two other sub-types described by Blaszczynski are characterized by conditions and histories that may be less effectively targeted by topiramate (i.e., impulsive, antisocial personality structure in the case of the Impulsive gamblers and irrational cognitions in the case of the Conditioned problem gambler). This population of gamblers, especially common among females, may report positive histories of substance abuse, anxiety and mood disorders, familial and childhood dysfunction, and familial gambling.

In an open-label study of topiramate with a sample of patients with post-traumatic stress disorder, an amelioration of dissociation and numbing was reported. These findings are also consistent with this medication's reported amnesic effects, and suggest that topiramate may reduce neural reactivity of problem gamblers that would otherwise increase the probability of engaging in gambling to self-regulate dysphoric emotional states.

The current study proposes to further evaluate the clinical efficacy of topiramate in a randomized, placebo-controlled clinical trial, the first study to do so. Interaction of the effects of the medication and gambling sub-type will be examined to determine whether the efficacy of topiramate is correlated with the specific biopsychosocial history of the gambler. An experimental trial of an acute dose of topiramate will run concurrently in order to identify cognitive-behavioural mechanisms that may mediate the clinical effects of topiramate on gambling-related behaviours evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* 19 - 65 years of age either gender
* plays electronic gaming machines (e.g. slot machine, video poker)
* meets DSM IV criteria for pathological gambling

Exclusion Criteria:

* females pregnant or breastfeeding at study entry
* females of childbearing age and physically able to conceive but not on oral contraceptives or patch, unwilling to take pregnancy self-test before each test session
* females taking oral contraceptives or patch but unwilling to use a barrier method of contraceptive during the course of the study
* occupation involving driving or operating heavy machinery
* BMI < 20
* hepatic dysfunction or hepatitis, as indicated by elevated INR, low serum albumin, or high bilirubin, or elevated AST, ALT, GGT (>1.5 times normal)
* clinical evidence of cirrhosis on examination
* renal insufficiency (creatinine >150)
* history of renal stones
* history of glaucoma
* current seizure disorder
* current use of digoxin
* current use of benzodiazepines
* alcohol consumption >14 drinks /week
* current use of anti-seizure medications (phenytoin, carbamazepine, valproic acid, primadone), antipsychotic medications (e.g., seroquel), carbonic anhydrase inhibitors (acetazolamide), metformin
* diagnosis of Axis I disorders, including psychoactive substances disorders (except nicotine)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Y-BOCS
CPGI

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Brands, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Grant JE, Kim SW, Potenza MN. Advances in the pharmacological treatment of pathological gambling. J Gambl Stud. 2003 Spring;19(1):85-109. doi: 10.1023/a:1021227214142. PMID 12635541
- [Background] Johnson BA, Ait-Daoud N, Akhtar FZ, Ma JZ. Oral topiramate reduces the consequences of drinking and improves the quality of life of alcohol-dependent individuals: a randomized controlled trial. Arch Gen Psychiatry. 2004 Sep;61(9):905-12. doi: 10.1001/archpsyc.61.9.905. PMID 15351769
- [Background] Dannon PN, Lowengrub K, Gonopolski Y, Musin E, Kotler M. Topiramate versus fluvoxamine in the treatment of pathological gambling: a randomized, blind-rater comparison study. Clin Neuropharmacol. 2005 Jan-Feb;28(1):6-10. doi: 10.1097/01.wnf.0000152623.46474.07. PMID 15711432
- [Background] Arnone D. Review of the use of Topiramate for treatment of psychiatric disorders. Ann Gen Psychiatry. 2005 Feb 16;4(1):5. doi: 10.1186/1744-859X-4-5. PMID 15845141
- [Background] Dannon PN. Topiramate for the treatment of kleptomania: a case series and review of the literature. Clin Neuropharmacol. 2003 Jan-Feb;26(1):1-4. doi: 10.1097/00002826-200301000-00001. PMID 12567156
- [Background] Blaszczynski A, Nower L. A pathways model of problem and pathological gambling. Addiction. 2002 May;97(5):487-99. doi: 10.1046/j.1360-0443.2002.00015.x. PMID 12033650
- [Background] Steel Z, Blaszczynski A. Impulsivity, personality disorders and pathological gambling severity. Addiction. 1998 Jun;93(6):895-905. doi: 10.1046/j.1360-0443.1998.93689511.x. PMID 9744125
- [Background] Petry NM, Steinberg KL; Women's Problem Gambling Research Center. Childhood maltreatment in male and female treatment-seeking pathological gamblers. Psychol Addict Behav. 2005 Jun;19(2):226-9. doi: 10.1037/0893-164X.19.2.226. PMID 16011396
- [Background] Berlant JL. Prospective open-label study of add-on and monotherapy topiramate in civilians with chronic nonhallucinatory posttraumatic stress disorder. BMC Psychiatry. 2004 Aug 18;4:24. doi: 10.1186/1471-244X-4-24. PMID 15315714
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research